CLINICAL TRIAL: NCT00516321
Title: Randomised, Placebo-controlled, Multi-centre Study to Assess the Efficacy and Safety of Eltrombopag in Thrombocytopenic Subjects With Hepatitis C Virus (HCV) Infection Who Are Otherwise Eligible to Initiate Antiviral Therapy (Peginterferon Alfa-2a Plus Ribavirin
Brief Title: Eltrombopag To Initiate And Maintain Interferon Antiviral Treatment To Subjects With Hepatitis C Related Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPL103922
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2012-08

CONDITIONS: Hepatitis C, Chronic
Keywords: thrombopoietin; hepatitis C; ribavirin; platelets; Hepatitis C-related thrombocytopenia; peginterferon alfa-2a
MeSH Terms: conditions — Hepatitis C, Chronic; Jacobs syndrome; Hepatitis C | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: eltrombopag — 25, 50, 75, 100 mg tablets taken once daily orally
Drug: placebo — matched placebo taken once daily orally

SUMMARY:
The purpose of this study is to assess the ability of eltrombopag to maintain a platelet count sufficient to facilitate initiation of antiviral therapy, to minimise antiviral therapy dose reductions and to avoid permanent discontinuation of antiviral therapy. The clinical benefit of eltrombopag will be measured by the proportion of subjects who are able to achieve a Sustained Virological Response (SVR).

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects, >18 years Evidence of chronic hepatitis C virus (HCV) infection Subjects who are appropriate candidates for peginterferon (pegIFN) and ribavirin antiviral therapy A platelet count of <75,000/mcL Haemoglobin >11.0g/dL for men or >10.0g/dL for women Absolute neutrophil count (ANC) >750/mm3 and no history of infections associated with neutropenia Creatinine clearance >50mL/minute All fertile males and females must use two forms of effective contraception between them during treatment and during the 24 weeks after treatment end Subject is able to understand, consent and comply with protocol requirements and instructions and is likely to complete the study as planned

Exclusion criteria:

Non-responders to previous treatment with pegIFN and ribavirin who failed to achieve a sustained virologic response (SVR) for reasons other than thrombocytopenia, despite an optimal course (dose and duration) of combination therapy with pegIFN and ribavirin Decompensated liver disease, e.g. Child-Pugh score >6 or history of ascites or hepatic encephalopathy or current evidence of ascites Known hypersensitivity, intolerance or allergy to interferon (IFN), ribavirin, eltrombopag or any of their ingredients Serious cardiac, cerebrovascular, or pulmonary disease that would preclude treatment with pegIFN and ribavirin

Subjects with a history of any one of the following:

Suicide attempt or hospitalisation for depression in the past 5 years Any current severe or poorly controlled psychiatric disorder

The following subjects are eligible for study participation, but must be assessed and followed (if recommended) by a mental health professional:

* Subjects who have had a severe or poorly controlled psychiatric disorder more than 6 months ago but less than 5 years ago
* Seizure disorder that has not been well controlled History of clinically significant bleeding from oesophageal or gastric varices Subjects with haemoglobinopathies, e.g. sickle cell anaemia, thalassemia major Any prior history of arterial or venous thrombosis AND two or more of the following risk factors: hereditary thrombophilic disorders (e.g. Factor V Leiden, antithrombin III (ATIII) deficiency, etc), hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension or cancer Pre-existing cardiac disease (New York Heart Association (NYHA) Grade III/IV), or arrhythmias known to involve the risk of thromboembolic events, or corrected QT interval (QTc) >450 msec Evidence of hepatocellular carcinoma Laboratory evidence of infection with human immunodeficiency virus (HIV) or active Hepatitis B Virus (HBV) infection Any disease condition associated with active bleeding or requiring anticoagulation with heparin or warfarin Therapy with any anti-neoplastic or immuno-modulatory treatment <6 months prior to the first dose of eltrombopag Subjects who have had a malignancy diagnosed and/or treated within the past 5 years, except for subjects with localised basal or squamous cell carcinoma treated by local excision or subjects with malignancies who have been adequately treated and, in the opinion of the oncologist, have an excellent chance of cancer-free survival Pregnant or nursing women Males with a female partner who is pregnant History of alcohol/drug abuse or dependence within 6 months of the study start (unless participating in a controlled rehabilitation programme) Treatment with an investigational drug or IFN within 30 days or 5 half-lives (whichever is longer) of the screening visit History of platelet clumping that prevents reliable measurement of platelet counts History of major organ transplantation with an existing functional graft Thyroid dysfunction not adequately controlled Subjects planning to have cataract surgery Evidence of portal vein thrombosis on abdominal imaging within 3 months of the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2007-10; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (166):
- United States (43):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Clemente, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Gainsville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Australia (7):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Brazil (2):
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- Canada (8):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Prague, Czechia
- France (8):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
- Germany (30):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Deggendorf, Bavaria
  - GSK Investigational Site, Hof/Saale, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Beeskow, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Leverkusen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Siegen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Pokfulam, Hong Kong
- India (3):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Mumbai
- Israel (5):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Safed
  - GSK Investigational Site, Tel Aviv
- Italy (10):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, San Giovanni Rotondo (FG), Apulia
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Palermo, Sicily
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, Lahore, Pakistan
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Wroclaw
- Puerto Rico (2):
  - GSK Investigational Site, Ponce, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Mosocow
  - GSK Investigational Site, Smolensk
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Martin
- South Korea (3):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (8):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, L'Hospitalet de Llobregat. Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Taiwan (4):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Thailand (4):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla
- Ukraine (3):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Vinnytsia
- United Kingdom (3):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, London
  - GSK Investigational Site, Plymouth

REFERENCES:
- [Derived] Saleh MI, Obeidat AR, Anter HA, Khanfar AA. Eltrombopag dose predictors in thrombocytopenic subjects with hepatitis C virus infection. Clin Exp Pharmacol Physiol. 2015 Oct;42(10):1030-5. doi: 10.1111/1440-1681.12451. PMID 26173631
- [Derived] Giannini EG, Afdhal NH, Sigal SH, Muir AJ, Reddy KR, Vijayaraghavan S, Elkashab M, Romero-Gomez M, Dusheiko GM, Iyengar M, Vasey SY, Campbell FM, Theodore D. Non-cirrhotic thrombocytopenic patients with hepatitis C virus: Characteristics and outcome of antiviral therapy. J Gastroenterol Hepatol. 2015 Aug;30(8):1301-8. doi: 10.1111/jgh.12942. PMID 25777337
- [Derived] Afdhal NH, Dusheiko GM, Giannini EG, Chen PJ, Han KH, Mohsin A, Rodriguez-Torres M, Rugina S, Bakulin I, Lawitz E, Shiffman ML, Tayyab GU, Poordad F, Kamel YM, Brainsky A, Geib J, Vasey SY, Patwardhan R, Campbell FM, Theodore D. Eltrombopag increases platelet numbers in thrombocytopenic patients with HCV infection and cirrhosis, allowing for effective antiviral therapy. Gastroenterology. 2014 Feb;146(2):442-52.e1. doi: 10.1053/j.gastro.2013.10.012. Epub 2013 Oct 12. PMID 24126097

RESULTS

PARTICIPANT FLOW:
Groups:
- Eltrombopag: OL Phase: Participants with a platelet count of <75 giga (10^9) cells per liter (Gi/L) initially received eltrombopag 25 milligrams (mg) once daily (QD) for 2 weeks. After 2 weeks, if the platelet count was <90 Gi/L, participants underwent dose escalation to 50 mg QD for 2 weeks. If platelet counts still remained <90 Gi/L, further dose escalations to 75 mg QD (up to 2 weeks) and 100 mg QD (up to a maximum of 3 weeks) were allowed. Participants who achieved platelet counts >=90 Gi/L during the OL Phase (maximum of up to 9 weeks) were eligible to enter the Double-blind (DB) Antiviral Treatment Phase, whereas those who failed to reach platelet counts >=90 Gi/L were discontinued from eltrombopag and had to attend the post-treatment follow-up visits.
- Placebo+Antiviral Therapy: DB Phase: Participants completing the OL Phase were administered matching placebo tablets QD in combination with antiviral therapy (peginterferon alfa-2a and ribavirin) for a duration of either 24 or 48 weeks (for participants with Genotype 2/3) or 48 weeks (for participants with Non-Genotype 2/3).
- Eltrombopag+Antiviral Therapy: DB Phase: Participants completing the OL Phase continued on the same dose of eltrombopag received in the OL Phase (dose that effectively raised platelets to >=90 Gi/L) in combination with antiviral therapy (peginterferon alfa-2a and ribavirin) for a duration of either 24 or 48 weeks (for participants with Genotype 2/3) or 48 weeks (for participants with Non-Genotype 2/3).
Period: Open-label (OL) Pre-Antiviral Treatment
Arm/Group | Eltrombopag: OL Phase | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Started | 715 | 0 | 0
Completed | 682 | 0 | 0
Not Completed | 33 | 0 | 0
Not completed — Lack of Efficacy | 11 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Investigator Discretion | 7 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Period: Double-blind (DB) Antiviral Treatment
Arm/Group | Eltrombopag: OL Phase | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Started | 0 | 232 | 450
Completed | 0 | 197 | 396
Not Completed | 0 | 35 | 54
Not completed — Lost to Follow-up | 0 | 12 | 22
Not completed — Withdrawal by Subject | 0 | 13 | 18
Not completed — Adverse Event | 0 | 8 | 13
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase | Total
Number analyzed (Participants) | 232 | 450 | 682
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected for the Intent-to-Treat (ITT) Population, which included all randomized participants in the Double-blind (DB) Phase of the study.
  Years
    Years | 51.4 (8.52) | 52.1 (8.35) | 51.9 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected for the Intent-to-Treat (ITT) Population, which included all randomized participants in the Double-blind (DB) Phase of the study.
  Participants
    Female | 73 | 186 | 259
    Male | 159 | 264 | 423
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study.
  participants
    African American/African Heritage | 6 | 12 | 18
    American Indian/Alaska Native | 3 | 2 | 5
    Central/South Asian Heritage | 14 | 39 | 53
    Japanese/East Asian Heritage/South East Asian | 43 | 68 | 111
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    White | 166 | 326 | 492
    Asian and White | 0 | 1 | 1
    Native Hawaiian/ Other Pacific Islander and White | 0 | 1 | 1
Number of participants categorized into the indicated genotype for Hepatitic C Virus (HCV) [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. The HCV is a small, enveloped, single-stranded, positive-sense ribonucleic acid (RNA) virus. There are seven major genotypes of HCV, which are indicated numerically from Genotype 1 to 7.
  participants
    Genotype 1 | 149 | 292 | 441
    Genotype 2 | 22 | 27 | 49
    Genotype 3 | 54 | 115 | 169
    Genotype 4 | 5 | 11 | 16
    Genotype 5 | 0 | 0 | 0
    Genotype 6 | 2 | 4 | 6
    Genotype 7 | 0 | 0 | 0
    Missing Data | 0 | 1 | 1
Number of participants categorized into the indicated Child-Pugh (CP) Class [Number; unit: participants] — The CP score (ranging from 5 to 15, with 5 being mild and 15 being severe), calculated based on total bilirubin, serum albumin, international normalized ratio, ascites, and hepatic encephalopathy, is used to assess the severity of liver disease. A CP score of 5-6 = Class A (mild); 7-9 = Class B (moderate); >=10 = Class C (severe).
  participants
    Class A | 217 | 424 | 641
    Class B | 15 | 25 | 40
    Class C | 0 | 0 | 0
    Missing Data | 0 | 1 | 1
Number of participants with or without previous interferon (IFN) use [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. Participants at Baseline were classified as not having used IFN previously (Naïve) or having used IFN previously (Experienced).
  participants
    Naïve | 152 | 307 | 459
    Experienced | 80 | 143 | 223
Number of participants with the indicated FibroTest/Acti Test (FibroSURE) score [Number; unit: participants] — FibroSURE is a noninvasive blood test that combines the quantitative results of 6 serum biochemical markers (α2-macroglobulin, haptoglobin, apolipoprotein A1, bilirubin, γ-glutamyl transpeptidase [GGT], and ALT) with a participant's age and gender to generate a measure of liver fibrosis/cirrhosis and necroinflammatory activity. It provides a numerical quantitative estimate of liver fibrosis ranging from 0.00 to 1.00, corresponding to the Metavir scoring system of stages F0 to F4 (F0, no fibrosis [F]; F1, portal F; F2, bridging F with few septa; F3, bridging F with many septa; F4=cirrhosis).
  participants
    Score: F0/F1/F2 | 23 | 37 | 60
    Score: F3/F4 | 185 | 354 | 539
    Missing | 24 | 59 | 83
Number of participants with normal or elevated Baseline values for Alanine Aminotransferase (ALT) [Number; unit: participants] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. The normal range of ALT is 0 to 48 International Units per Liter (IU/L).
  participants
    Normal | 54 | 103 | 157
    Elevated | 178 | 347 | 525
Baseline HCV Ribonucleic Acid (RNA) [Mean (Standard Deviation); unit: International Units per milliliter] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. HCV RNA was assessed at baseline of the DB Phase. Data are missing for one participant in the Eltrombopag+Antiviral Therapy treatment group.
  International Units per milliliter | 1880278.4 (3395777.02) | 1870562.1 (3080918.03) | 1873862.8 (3188864.74)
Baseline Platelet Count [Mean (Standard Deviation); unit: Giga (10^9) cells per liter (Gi/L)] — Baseline characteristics were collected for the ITT Population, which included all randomized participants in the DB Phase of the study. Platelet count eligibility was confirmed at the Baseline visit, prior to administration of eltrombopag, and was defined as the average of the screening and baseline counts, which must be <75 Gi/L.
  Giga (10^9) cells per liter (Gi/L) | 57.40 (12.890) | 56.87 (13.603) | 57.05 (13.357)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR) in the Double-blind (DB) Antiviral Treatment Phase
Description: Participants with SVR were defined as those with undetectable Hepatitis C Virus (HCV) ribonucleic acid (RNA) at 24 weeks post-completion of the treatment period of the DB Phase.
Time Frame: From Baseline up to Week 48 or Week 72 (for participants with Genotype 2/3) or up to Week 72 (for participants with Non-Genotype 2/3)
Population: Intent-to-Treat (ITT) Population: all participants randomized in the DB Phase
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants | 33 | 104
Statistical Analysis 1: Comparison: Placebo+Antiviral Therapy: DB Phase vs Eltrombopag+Antiviral Therapy: DB Phase; Test type: Superiority or Other; p = 0.0064, Cochran-Mantel-Haenszel — Stratified Cochran-Mantel-Haenszel (CMH) chi-square test adjusted for the randomization strata; Percentage difference in SVR = 7.9, 95% CI 2-sided [2.4 to 13.4] — The estimated value reflects the percentage of participants with SVR in the eltrombopag group minus the percentage of participants with SVR in the placebo group. Adjusted for the actual strata: HCV genotype, baseline platelet count, and HCV RNA

2. Secondary Outcome: Number of Participants Whose Platelet Count Increased From a Baseline Count of <75 Gi/L to a Count Greater Than or Equal to (>=) 90 Giga (10^9) Cells Per Liter (Gi/L) During the Open-label (OL) Pre-Antiviral Treatment Phase
Description: Participants were assessed for a shift from a baseline platelet count of <75 Gi/L to a count >=90 Gi/L during the OL Phase (up to 9 weeks). Local laboratories were used for platelet function tests. Platelet counts were measured by blood draw.
Time Frame: From Baseline up to Week 9 in the OL Phase
Population: Safety Population: all participants who had received study drug in the OL Phase
Measure: Number; unit: participants
Arm/Group | Eltrombopag: OL Phase
Number analyzed (Participants) | 715
participants | 691

3. Secondary Outcome: Number of Participants Receiving the Indicated Doses of Eltrombopag in the OL Phase Who Initiated Antiviral Therapy (Peginterferon Alfa-2a and Ribavirin) in the DB Phase
Description: In the OL Phase, participants initially received the lowest dose of eltrombopag (25 mg QD) for 2 weeks. If after this time the platelet count was <90 Gi/L, participants underwent sequential dose escalation to the next highest dose (50 mg QD for up to 2 weeks), with further dose escalations to 75 mg QD (up to 2 weeks) and 100 mg QD (up to a maximum of 3 weeks) if platelet counts remained <90 Gi/L. Participants who achieved platelet count >=90 Gi/L on any of the eltrombopag doses in the OL Phase initiated antiviral therapy in the DB Phase.
Time Frame: From Baseline up to Week 9 in the OL Phase
Population: Safety Population. Participants with a platelet count >=90 Gi/L and who initiated antiviral therapy during the DB Phase were analyzed.
Measure: Number; unit: participants
Arm/Group | Eltrombopag: OL Phase
Number analyzed (Participants) | 680
participants
  25 mg | 451
  50 mg | 176
  75 mg | 39
  100 mg | 14

4. Secondary Outcome: Median Platelet Count at the Indicated Time Points During the OL Phase
Description: Blood taken from peripheral blood vessels was used for the measurement of platelet counts. The Last On Treatment assessment refers to the actual last treatment assessment, not necessarily to the End of Treatment assessment entered by the Investigator.
Time Frame: OL Phase: Baseline; Day 1; Weeks 1, 2, 3, 4, 5, 6, 7, 8, and 9; Antiviral Baseline (up to Week 10); End of Treatment (up to Week 48); 4-week Follow-up (FU) (up to Week 62); 12-week FU (up to Week 70); and 24-week FU (up to Week 82)
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Eltrombopag: OL Phase
Number analyzed (Participants) | 712
Gi/L
  Baseline, n=712 | 59.00 [3.00 to 98.34]
  Day 1, n=620 | 59.00 [5.00 to 108.00]
  Week 1, n=703 | 77.00 [7.00 to 226.00]
  Week 2, n=426 | 89.00 [11.00 to 389.58]
  Week 3, n=179 | 83.00 [11.00 to 335.00]
  Week 4, n=98 | 83.00 [12.00 to 310.00]
  Week 5, n=56 | 77.00 [16.00 to 379.00]
  Week 6, n=35 | 79.00 [24.00 to 436.00]
  Week 7, n=29 | 77.00 [30.00 to 187.90]
  Week 8, n=18 | 83.00 [37.00 to 135.00]
  Week 9, n=7 | 70.00 [38.00 to 113.00]
  Antiviral Baseline, n=48 | 130.00 [90.00 to 291.00]
  End of Treatment/Withdrawal, n=18 | 63.00 [6.00 to 331.97]
  Last on Treatment, n=30 | 75.00 [6.00 to 249.56]
  4 Week Follow-Up, n=15 | 44.00 [4.00 to 248.85]
  12 Week Follow-Up, n=16 | 38.00 [19.00 to 86.00]
  24 Week Follow-Up, n=15 | 38.00 [9.00 to 79.00]

5. Secondary Outcome: Median Platelet Count at the Indicated Time Points During the DB Phase
Description: Blood taken from peripheral blood vessels was used for the measurement of platelet counts.
Time Frame: DB Phase: Baseline; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44; End of Treatment (up to Week 48); 4-week Follow-up (FU) (up to Week 52); 12-week FU (up to Week 60); and 24-week FU (up to Week 72)
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed. The Last On Treatment assessment refers to the actual last treatment assessment, not necessarily to the End of Treatment assessment entered by the Investigator.
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 447
Gi/L
  Baseline, n=208, 387 | 128.00 [84.00 to 521.00] | 133.00 [64.00 to 509.00]
  Week 1, n=227, 443 | 112.00 [30.00 to 398.00] | 115.00 [31.00 to 502.00]
  Week 2, n=227, 438 | 79.00 [25.00 to 297.00] | 111.00 [36.00 to 596.00]
  Week 4, n=218, 430 | 43.50 [17.00 to 275.00] | 90.00 [5.00 to 430.00]
  Week 6, n=197, 423 | 40.00 [12.00 to 261.00] | 89.00 [22.00 to 315.00]
  Week 8, n=189, 414 | 41.00 [15.00 to 320.00] | 86.00 [22.00 to 249.00]
  Week 12, n=165, 404 | 44.00 [16.00 to 284.00] | 91.50 [25.00 to 298.00]
  Week 16, n=141, 377 | 43.00 [16.00 to 280.00] | 93.00 [26.00 to 376.00]
  Week 20, n=135, 363 | 44.00 [18.00 to 325.00] | 89.00 [25.00 to 339.00]
  Week 24, n=89, 248 | 43.00 [21.00 to 333.00] | 92.00 [18.00 to 276.00]
  Week 28, n=73, 202 | 45.00 [22.00 to 345.00] | 89.50 [17.00 to 207.00]
  Week 32, n=69, 183 | 44.40 [24.00 to 338.00] | 91.00 [21.00 to 406.00]
  Week 36, n=68, 173 | 44.50 [16.00 to 315.00] | 91.00 [21.00 to 209.00]
  Week 40, n=64, 169 | 44.00 [22.00 to 276.00] | 93.00 [30.00 to 226.00]
  Week 44, n=65, 168 | 48.00 [22.00 to 320.00] | 93.50 [27.00 to 238.00]
  End of Treatment/Withdrawal, n=212, 419 | 40.00 [8.00 to 318.00] | 90.00 [5.00 to 420.00]
  Last on Treatment, n=232, 447 | 40.00 [8.00 to 318.00] | 90.00 [5.00 to 420.00]
  4 Week Follow-Up, n=205, 400 | 54.00 [5.00 to 358.00] | 82.00 [5.00 to 304.00]
  12 Week Follow-Up, n=196, 396 | 56.00 [8.00 to 311.00] | 67.00 [1.00 to 350.00]
  24 Week Follow-Up, n=193, 391 | 56.00 [9.00 to 433.00] | 60.00 [7.00 to 340.00]

6. Secondary Outcome: Number of Participants in the Indicated Categories for Minimum Platelet Count With Antiviral Therapy During the DB Phase
Description: The minimum platelet count with antiviral therapy was categorized as follows: <25 Gi/L; >=25 to <50 Gi/L; >=50 to <90 Gi/L; >=90 to <150 Gi/L; >=150 Gi/L to <200 Gi/L; >=200 Gi/L to <400 Gi/L; and >=400 Gi/L.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants
  <25 Gi/L | 63 | 12
  >=25 to <50 Gi/L | 135 | 125
  >=50 to <90 Gi/L | 19 | 245
  >=90 to <150 Gi/L | 11 | 58
  >=150 to <200 Gi/L | 2 | 6
  >=200 to <400 Gi/L | 2 | 1
  >=400 Gi/L | 0 | 0
  Missing | 0 | 3

7. Secondary Outcome: Number of Participants With Rapid Virological Response (RVR) and Extended RVR (eRVR) During the DB Phase
Description: RVR is defined as the absence of detectable HCV RNA after 4 weeks of antiviral treatment. eRVR is defined as the absence of detectable HCV RNA after 4 weeks of antiviral treatment that persisted through Week 12.
Time Frame: From Baseline up to Week 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants
  RVR | 39 | 73
  eRVR | 28 | 68

8. Secondary Outcome: Number of Participants With Early Virological Response (EVR) and Complete EVR (cEVR) During the DB Phase
Description: EVR is defined as a clinically significant reduction from Baseline in HCV RNA (>=2 log10 decrease in HCV RNA or undetectable HCV RNA) after 12 weeks of antiviral treatment. cEVR, a subset of EVR, is defined exclusively as undetectable HCV RNA after 12 weeks of antiviral treatment.
Time Frame: From Baseline up to Week 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants
  EVR | 115 | 297
  cEVR | 60 | 187

9. Secondary Outcome: Number of Participants With End of Treatment Response (ETR) and Sustained Virological Response at Week 12 of Follow-up (SVR12) During the DB Phase
Description: ETR is defined as the absence of detectable HCV RNA at the end of antiviral treatment. SVR12 is defined as the absence of detectable HCV RNA at the end of antiviral treatment and the 12-week follow-up assessment.
Time Frame: From Baseline up to Week 36 or Week 60 (for participants with Genotype 2/3) or up to Week 60 (for participants with Non-Genotype 2/3)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants
  ETR | 86 | 214
  SVR12 | 36 | 347

10. Secondary Outcome: Number of Participants in the Indicated Categories for Antiviral Therapy Dose Reductions in the DB Phase
Description: Participants were assigned a score equal to the number of times their dose of antiviral therapy (peginterferon or ribavirin) was reduced (0=no dose reductions [DRs]; 1=one DR; 2=two DRs; 3=three DRs; >3=more than three DRs). Where possible, every effort was made to maintain the recommended dose of antiviral therapy for the treatment duration in the DB Phase. However, where dose modification of antiviral therapy was required due to safety concerns, it was performed by the Investigator as per the region-specific product labels of peginterferon and ribavirin.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants
  0 | 65 | 195
  1 | 57 | 93
  2 | 55 | 56
  3 | 26 | 49
  >3 | 29 | 57

11. Secondary Outcome: Time to First Dose Reduction of Peginterferon Alfa-2a and Ribavirin Therapy in the DB Phase
Description: Time to first dose reduction was calculated as the time period from the first dose to the first dose reduction.
Time Frame: as for outcome 1
Population: ITT Population. Only those participants with dose reductions were analyzed.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 163 | 193
weeks
  Peginterferon alfa-2a dose reduction, n=163, 193 | 5.81 (5.304) | 9.04 (9.371)
  Ribavirin dose reduction, n=63, 162 | 11.16 (9.219) | 12.58 (9.830)

12. Secondary Outcome: Number of Participants With the Indicated Levels of Peginterferon Dose Reductions in the DB Phase
Description: The assigned dose in the DB Phase of peginterferon alfa-2a was 180 micrograms (mcg). For peginterferon dose modification, downward adjustments in one level increments was considered. The lowest dose of peginterferon alfa-2a that was allowed to be administered was 45 mcg. Where dose adjustment was required for moderate to severe adverse reactions (clinical and/or laboratory), an initial dose reduction to 135 mcg was generally adequate. In some cases, a dose reduction to 90 mcg or 45mcg was necessary. Dose increases toward the original dose were considered when the adverse reaction was resolved.
Time Frame: as for outcome 1
Population: ITT Population. One participant could have had more than one dose reduction.
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants
  180 to 135 mcg | 73 | 121
  180 to 90 mcg | 94 | 82
  180 to 45 mcg | 2 | 0
  135 to 90 mcg | 55 | 64
  135 to 45 mcg | 2 | 0
  90 to 45 mcg | 18 | 12

13. Secondary Outcome: Number of Participants Who Prematurely Discontinued Antiviral Therapy in the DB Phase
Description: The following participants were considered to have discontinued from antiviral therapy: participants who were lost to follow-up; participants who withdrew for any reason; participants who died; participants who otherwise did not complete their planned course of antiviral therapy for any reason. The planned duration of antiviral therapy was 48 weeks for participants with Non-Genotype 2/3 and 24 or 48 weeks for participants with Genotype 2/3.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 450
participants | 129 | 184

14. Secondary Outcome: Number of Participants (Par.) Categorized as Responders (R) and Non-responders (NR) for SVR and RVR to Antiviral Therapy in the Indicated Variants of Interleukin 28B (IL28B) (or Interferon, Lambda 3) During the DB Phase
Description: There are two genetic variants (rs12979860 and rs8099917) mapping near IL28B associated with both interferon-induced SVR and spontaneous HCV clearance. Genotyping of the IL28B polymorphisms (rs12979860 and rs8099917) was conducted. IL28B genotype distribution by response to antiviral therapy (SVR and RVR) for both treatment arms was assessed. The effect of genotype was tested by comparing participants that carried 2 copies of the IL28B favorable response allele versus the others (recessive model). Genotypes at rs12979860 were coded as: CC=1, CT or TT=0; rs8099917 was coded as TT=1, GT or GG=0.
Time Frame: as for outcome 1
Population: Pharmacogenetic (PGx) Sub-Population: participants enrolled in this study who provided written informed consent for PGx research with a blood sample for genotyping and who were successfully genotyped for at least one of the two genetic markers under study
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 99 | 181
participants
  SVR, rs12979860 (CC), R; n=12, 36 | 5 | 18
  SVR, rs12979860 (CC), NR; n=99, 168 | 21 | 38
  SVR, rs12979860 (CT), R; n=12, 36 | 6 | 17
  SVR, rs12979860 (CT), NR; n=99, 168 | 63 | 95
  SVR, rs12979860 (TT), R; n=12, 36 | 1 | 1
  SVR, rs12979860 (TT), NR; n=99, 168 | 15 | 35
  SVR, rs8099917 (TT), R; n=12, 36 | 7 | 26
  SVR, rs8099917 (TT), NR; n=99, 166 | 50 | 70
  SVR, rs8099917 (GT), R; n=12, 36 | 4 | 9
  SVR, rs8099917 (GT), NR; n=99, 166 | 42 | 75
  SVR, rs8099917 (GG), R; n=12, 36 | 1 | 1
  SVR, rs8099917 (GG), NR; n=99, 166 | 7 | 21
  RVR, rs12979860 (CC), R; n=16, 23 | 7 | 12
  RVR, rs12979860 (CC), NR; n=95, 181 | 19 | 44
  RVR, rs12979860 (CT), R; n=16, 23 | 7 | 10
  RVR, rs12979860 (CT), NR; n=95, 181 | 62 | 102
  RVR, rs12979860 (TT), R; n=16, 23 | 2 | 1
  RVR, rs12979860 (TT), NR; n=95, 181 | 14 | 35
  RVR, rs8099917 (TT), R, n=16, 23 | 10 | 14
  RVR, rs8099917 (TT), NR; n=95, 179 | 47 | 82
  RVR, rs8099917 (GT), R; n=16, 23 | 4 | 9
  RVR, rs8099917 (GT), NR; n=95, 179 | 42 | 75
  RVR, rs8099917 (GG), R; n=16, 23 | 2 | 0
  RVR, rs8099917 (GG), NR; n=95, 179 | 6 | 22

15. Secondary Outcome: Number of Par. With the Indicated Shift From Baseline (BL) in Severity Grades for Clinical Chemistry Parameters (Calcium, Glucose [Glu.], Potassium [Pot.], and Sodium [Sod.]), Per Division of Acquired Immunodeficiency Syndrome (DAIDS) During the DB Phase
Description: Blood samples for the assessment of clinical chemistry parameters were taken at intervals throughout the study. Participants with the worst-case shift from BL during the DB Phase are reported, per severity grades by DAIDS, for levels of calcium (low=hypocalcemia; high=hypercalcemia), glu. (low=hypoglycemia; high=hyperglycemia), pot. (low=hypokalemia; high=hyperkalemia), and sod. (low=hyponatremia; high=hypernatremia). Per the DAIDS toxicity table, the grade ranges for each parameter are as follows: Grade (G) 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: as for outcome 1
Population: Safety DB Population: all randomized participants who had received study drug in the DB Phase
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 449
participants
  Calcium (hypocalcemia), Any Grade Increase | 173 | 343
  Calcium (hypocalcemia), Increase to G1 | 127 | 211
  Calcium (hypocalcemia), Increase to G2 | 45 | 126
  Calcium (hypocalcemia), Increase to G3 | 1 | 4
  Calcium (hypocalcemia), Increase to G4 | 0 | 2
  Calcium (hypercalcemia), Any Grade Increase | 1 | 5
  Calcium (hypercalcemia), Increase to G1 | 0 | 4
  Calcium (hypercalcemia), Increase to G2 | 1 | 1
  Calcium (hypercalcemia), Increase to G3 | 0 | 0
  Calcium (hypercalcemia), Increase to G4 | 0 | 0
  Glu. (hypoglycemia), Any Grade Increase | 23 | 58
  Glu. (hypoglycemia), Increase to G1 | 14 | 30
  Glu. (hypoglycemia), Increase to G2 | 6 | 22
  Glu. (hypoglycemia), Increase to G3 | 1 | 4
  Glu. (hypoglycemia), Increase to G4 | 2 | 2
  Glu. (hyperglycemia), Any Grade Increase | 111 | 239
  Glu. (hyperglycemia), Increase to G1 | 28 | 61
  Glu. (hyperglycemia), Increase to G2 | 62 | 148
  Glu. (hyperglycemia), Increase to G3 | 19 | 29
  Glu. (hyperglycemia), Increase to G4 | 2 | 1
  Pot. (hyperkalemia), Any Grade Increase | 6 | 10
  Pot. (hyperkalemia), Increase to G1 | 2 | 6
  Pot. (hyperkalemia), Increase to G2 | 1 | 2
  Pot. (hyperkalemia), Increase to G3 | 1 | 1
  Pot. (hyperkalemia), Increase to G4 | 2 | 1
  Pot. (hypokalemia), Any Grade Increase | 33 | 58
  Pot. (hypokalemia), Increase to G1 | 29 | 53
  Pot. (hypokalemia), Increase to G2 | 4 | 5
  Pot. (hypokalemia), Increase to G3 | 0 | 0
  Pot. (hypokalemia), Increase to G4 | 0 | 0
  Sod. (hypernatremia), Any Grade Increase | 9 | 12
  Sod. (hypernatremia), Increase to G1 | 9 | 11
  Sod. (hypernatremia), Increase to G2 | 0 | 0
  Sod. (hypernatremia), Increase to G3 | 0 | 0
  Sod. (hypernatremia), Increase to G4 | 0 | 1
  Sod. (hyponatremia), Any Grade Increase | 65 | 151
  Sod. (hyponatremia), Increase to G1 | 62 | 134
  Sod. (hyponatremia), Increase to G2 | 3 | 11
  Sod. (hyponatremia), Increase to G3 | 0 | 3
  Sod. (hyponatremia), Increase to G4 | 0 | 3

16. Secondary Outcome: Number of Participants With the Indicated Shifts From BL in Severity Grades for for Hematology Parameters (Hemoglobin, Lymphocytes [Lym.], Total Neutrophils [Tot Neu.], and White Blood Cells [WBC]), Per DAIDS During the DB Phase
Description: Blood samples for the assessment of hematology parameters were taken at intervals throughout the study. Participants with the worst-case shift from BL during the DB Phase are reported, per severity grades by DAIDS, for levels of hemoglobin (low=anemia), lymphocytes (low=lymphocytopenia), total neutrophils (low=neutropenia), and white blood cells (low=leukocytopenia). Per the DAIDS toxicity table, grade ranges for each parameter are as follows: Grade (G) 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: as for outcome 1
Population: Safety DB Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 449
participants
  Hemoglobin (anemia), Any Grade Increase | 148 | 324
  Hemoglobin (anemia), Increase to G1 | 45 | 91
  Hemoglobin (anemia), Increase to G2 | 63 | 128
  Hemoglobin (anemia), Increase to G3 | 37 | 98
  Hemoglobin (anemia), Increase to G4 | 3 | 7
  Lym. (lymphocytopenia), Any Grade Increase | 123 | 300
  Lym. (lymphocytopenia), Increase to G1 | 16 | 26
  Lym. (lymphocytopenia), Increase to G2 | 28 | 50
  Lym. (lymphocytopenia), Increase to G3 | 43 | 96
  Lym. (lymphocytopenia), Increase to G4 | 36 | 128
  Tot Neu. (neutropenia), Any Grade Increase | 196 | 394
  Tot Neu. (neutropenia), Increase to G1 | 32 | 90
  Tot Neu. (neutropenia), Increase to G2 | 39 | 104
  Tot Neu. (neutropenia), Increase to G3 | 80 | 129
  Tot Neu. (neutropenia), Increase to G4 | 45 | 71
  WBC (leukocytopenia), Any Grade Increase | 187 | 376
  WBC (leukocytopenia), Increase to G1 | 51 | 94
  WBC (leukocytopenia), Increase to G2 | 59 | 142
  WBC (leukocytopenia), Increase to G3 | 68 | 117
  WBC (leukocytopenia), Increase to G4 | 9 | 23

17. Secondary Outcome: Number of Participants in the Indicated Categories for Cataract Event During the DB Phase, Per Clinical Events Committee (CEC) Adjudication During the DB Phase
Description: Ophthalmic (pertaining to eye) assessments were performed during the study. A cataract event is defined as an event ascertained to be a cataract (opacity or cloudiness of the lens of the eye, causing impairment of vision) by at least one of the CEC members (comprised of expert ophthalmologists who provided objective medical review of the blinded ophthalmic data). Per the CEC, cataract events were categorized as: (1) Cataract Progression (CP; progression of cataracts present at BL); and (2) Incident Cataract (IC; development of new cataracts). One eye=unilateral; both eyes=bilateral.
Time Frame: as for outcome 1
Population: Safety DB Population
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 232 | 449
participants
  Unilateral CP, Genotype 2/3 | 1 | 2
  Unilateral CP, Non-genotype 2/3 | 2 | 3
  Unilateral CP, Missing genotype | 0 | 1
  Bilateral CP, Genotype 2/3 | 1 | 6
  Bilateral CP, Non-genotype 2/3 | 0 | 9
  Unilateral IP, Genotype 2/3 | 0 | 1
  Unilateral IP, Non-genotype 2/3 | 2 | 6
  Bilateral IP, Genotype 2/3 | 2 | 2
  Bilateral IP, Non-genotype 2/3 | 0 | 8

18. Secondary Outcome: Number of Participants Assessed as Normal and Abnormal (Clinically Significant [CS] and Not Clinically Significant [NCS]) for 12-lead Electrocardiogram (ECG) at the Indicated Time Points During the DB Phase
Description: Duplicate 12-lead ECGs were required at Screening/BL, Antiviral BL, and at 12 weekly intervals during the study. The investigator assigned an ECG status of normal, abnormal, CS, or NCS; a status of "abnormal" alone indicates that the investigator did not determine if ECG was CS or NCS. Normal, all ECG parameters within accepted normal ranges. Abnormal, ECG finding(s) outside of normal ranges. CS, ECG with a CS abnormality that meets exclusion criteria. NCS, ECG with an abnormality not CS or meeting exclusion criteria, per Investigator, based on reasonable standards of clinical judgment.
Time Frame: DB Phase: Antiviral BL (up to Week 10); End of Treatment (up to Week 52); and 24-week FU (up to Week 72)
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed. Worst ECG post-BL is the worst ECG assessment reported for a participant at a post-BL assessment and could be Normal, Abnormal - NCS, Abnormal - CS, or Abnormal (NCS or CS not given).
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 229 | 447
participants
  Antiviral BL, Normal, n=219, 423 | 149 | 278
  Antiviral BL, Abnormal - NCS, n=219, 423 | 53 | 108
  Antiviral BL, Abnormal - CS, n=219, 423 | 17 | 37
  End of Treatment, Normal, n=198, 384 | 139 | 251
  End of Treatment, Abnormal - NCS, n=198, 384 | 50 | 108
  End of Treatment, Abnormal - CS, n=198, 384 | 9 | 24
  End of Treatment, Abnormal, n=198, 384 | 0 | 1
  24-week FU, Normal, n=186, 368 | 120 | 235
  24-week FU, Abnormal - NCS, n=186, 368 | 53 | 106
  24-week FU, Abnormal - CS, n=186, 368 | 13 | 27
  Worst ECG post-BL, Normal, n=229, 447 | 105 | 188
  Worst ECG post-BL, Abnormal - NCS, n=229, 447 | 87 | 186
  Worst ECG post-BL, Abnormal - CS, n=229, 447 | 37 | 72
  Worst ECG post-BL, Abnormal, n=229, 447 | 0 | 1

19. Secondary Outcome: Number of Participants With CS and NCS Change From Baseline for 12-lead ECG at the Indicated Time Points During the DB Phase
Description: Duplicate 12-lead ECGs were required at Screening/BL, Antiviral BL, and at 12 weekly intervals during the study. The number of participants with a CS or a NCS change from baseline in ECG status was reported, as determined by the Investigator based on a reasonable standard of clinical judgment. "Not applicable" indicates that information was not provided by the investigator on whether the change from baseline ECG was CS or NCS.
Time Frame: End of Treatment (up to Week 52); and 24-week FU (up to Week 72)
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 198 | 383
participants
  End of Treatment, CS change from BL, n=198, 383 | 2 | 5
  End of Treatment, NCS change from BL, n=198, 383 | 196 | 377
  End of Treatment, Not applicable, n=198, 383 | 0 | 1
  24-week FU, CS change from BL, n=186, 369 | 1 | 8
  24-week FU, NCS change from BL, n=186, 369 | 185 | 361

20. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points During the DB Phase
Description: Participant's blood pressure was measured at the indicated time points during the study. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic blood pressure is a measure of blood pressure while the heart is relaxed. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 231 | 444
Millimeters of mercury (mmHg)
  SBP, Week 1, n=231, 443 | -3.3 (13.66) | -2.7 (13.48)
  SBP, Week 2, n=227, 437 | -5.0 (13.75) | -3.2 (14.05)
  SBP, Week 4, n=218, 429 | -6.1 (13.61) | -3.7 (13.63)
  SBP, Week 6, n=196, 420 | -4.3 (14.00) | -3.9 (13.86)
  SBP, Week 8, n=190, 416 | -3.6 (14.04) | -3.9 (14.15)
  SBP, Week 12, n=165, 405 | -4.0 (13.17) | -3.6 (14.07)
  SBP, Week 16, n=140, 376 | -4.2 (13.69) | -3.8 (13.88)
  SBP, Week 20, n=135, 363 | -4.1 (15.09) | -3.2 (14.84)
  SBP, Week 24, n=88, 249 | -3.7 (15.88) | -2.9 (15.88)
  SBP, Week 28, n=74, 202 | -3.0 (12.79) | -3.3 (16.62)
  SBP, Week 32, n=68, 183 | -3.1 (11.95) | -2.6 (16.12)
  SBP, Week 36, n=68, 175 | -2.4 (13.73) | -3.0 (16.43)
  SBP, Week 40, n=64, 169 | -2.7 (11.95) | -3.4 (16.47)
  SBP, Week 44, n=64, 166 | -2.5 (12.98) | -3.8 (16.76)
  SBP, End of Treatment, n=213, 420 | -3.8 (14.94) | -3.1 (15.65)
  SBP, 4-week FU, n=204, 402 | -0.7 (13.95) | -1.2 (16.23)
  SBP, 12-week FU, n=198, 401 | -0.4 (14.24) | -0.7 (15.68)
  SBP, 24-week FU, n=197, 394 | -0.1 (14.04) | 0.1 (16.02)
  DBP, Week 1, n=231, 443 | -1.3 (9.57) | -1.5 (9.21)
  DBP, Week 2, n=227, 437 | -2.6 (10.05) | -1.8 (9.11)
  DBP, Week 4, n=218, 429 | -3.2 (10.01) | -2.3 (10.12)
  DBP, Week 6, n=196, 420 | -1.9 (9.13) | -3.1 (9.69)
  DBP, Week 8, n=190, 416 | -2.7 (9.67) | -2.6 (10.03)
  DBP, Week 12, n=165, 405 | -3.0 (9.92) | -2.8 (10.05)
  DBP, Week 16, n=140, 376 | -2.4 (9.19) | -3.1 (10.01)
  DBP, Week 20, n=135, 363 | -3.5 (10.04) | -2.4 (9.59)
  DBP, Week 24, n=88, 249 | -2.4 (10.60) | -2.9 (9.95)
  DBP, Week 28, n=74, 202 | -3.7 (10.32) | -3.0 (10.43)
  DBP, Week 32, n=68, 183 | -1.7 (10.93) | -2.5 (9.99)
  DBP, Week 36, n=68, 175 | -1.5 (11.51) | -3.1 (9.84)
  DBP, Week 40, n=64, 169 | -2.7 (10.65) | -2.9 (10.99)
  DBP, Week 44, n=64, 166 | -2.8 (10.96) | -3.2 (10.54)
  DBP, End of Treatment, n=213, 420 | -2.8 (10.07) | -2.8 (10.26)
  DBP, 4-week FU, n=204, 402 | -1.8 (9.30) | -1.2 (10.67)
  DBP, 12-week FU, n=198, 401 | -1.4 (10.48) | -0.9 (10.09)
  DBP, 24-week FU, n=197, 394 | -0.6 (9.90) | -0.3 (9.97)

21. Secondary Outcome: Mean Change From Baseline in Heart Rate at the Indicated Time Points During the DB Phase
Description: Heart rate was measured in participants at the indicated time points. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 231 | 443
beats per minute
  Week 1, n=231, 440 | 0.6 (8.99) | 0.9 (8.50)
  Week 2, n=227, 435 | 1.1 (9.31) | 2.3 (9.16)
  Week 4, n=217, 428 | 1.7 (9.83) | 2.7 (9.01)
  Week 6, n=195, 419 | 2.3 (11.74) | 2.9 (8.88)
  Week 8, n=190, 414 | 2.3 (10.27) | 3.6 (9.98)
  Week 12, n=164, 404 | 3.8 (11.30) | 4.1 (9.93)
  Week 16, n=140, 375 | 4.7 (11.81) | 4.2 (9.87)
  Week 20, n=135, 363 | 3.4 (11.05) | 4.8 (9.73)
  Week 24, n=88, 248 | 4.8 (11.34) | 4.7 (10.91)
  Week 28, n=73, 200 | 4.6 (10.29) | 4.5 (9.75)
  Week 32, n=68, 182 | 6.1 (10.48) | 5.5 (10.46)
  Week 36, n=68, 174 | 5.5 (11.55) | 4.1 (11.84)
  Week 40, n=64, 166 | 5.8 (9.33) | 5.0 (10.32)
  Week 44, n=64, 166 | 5.3 (11.30) | 5.5 (9.94)
  End of Treatment, n=212, 419 | 2.9 (10.54) | 4.3 (10.84)
  4-week FU, n=204, 397 | 2.7 (11.47) | 3.5 (10.38)
  12-week FU, n=197, 400 | 0.5 (11.23) | 1.7 (10.40)
  24-week FU, n=197, 393 | 0.1 (11.61) | 0.5 (10.34)

22. Secondary Outcome: Mean Change From Baseline in Weight at the Indicated Time Points During the DB Phase
Description: The weight of participants was recorded at the indicated time points. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 230 | 443
Kilograms (kg)
  Week 1, n=230, 443 | -0.5 (1.83) | -0.6 (1.76)
  Week 2, n=227, 439 | -0.7 (1.95) | -0.7 (1.87)
  Week 4, n=218, 430 | -0.8 (2.16) | -1.0 (2.39)
  Week 6, n=198, 421 | -1.0 (2.30) | -1.2 (2.33)
  Week 8, n=191, 416 | -1.2 (2.63) | -1.7 (2.68)
  Week 12, n=165, 404 | -1.4 (3.27) | -2.3 (3.15)
  Week 16, n=139, 377 | -1.8 (3.15) | -2.8 (3.19)
  Week 20, n=135, 364 | -2.0 (3.74) | -3.3 (3.62)
  Week 24, n=88, 249 | -1.7 (3.59) | -4.1 (3.88)
  Week 28, n=74, 202 | -2.5 (4.79) | -4.4 (3.96)
  Week 32, n=69, 184 | -1.8 (3.70) | -4.2 (4.01)
  Week 36, n=68, 175 | -1.9 (3.81) | -4.4 (4.07)
  Week 40, n=64, 169 | -1.8 (4.10) | -4.5 (4.30)
  Week 44, n=65, 166 | -2.0 (4.40) | -4.7 (4.35)
  End of Treatment, n=214, 419 | -2.0 (3.88) | -4.2 (4.65)
  4-week FU, n=204, 404 | -2.0 (3.95) | -3.7 (4.68)
  12-week FU, n=198, 401 | -1.4 (4.51) | -2.9 (5.07)
  24-week FU, n=197, 393 | -0.7 (5.32) | -1.8 (5.14)

23. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI) at the Indicated Time Points During the DB Phase
Description: The BMI for participants was calculated at the indicated time points as body weight in kilograms divided by height in meters squared. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: as for outcome 5
Population: Safety DB Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms per meters squared (kg/m^2)
Arm/Group | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Number analyzed (Participants) | 228 | 440
Kilograms per meters squared (kg/m^2)
  Week 1, n=228, 440 | -0.2 (0.61) | -0.2 (0.61)
  Week 2, n=225, 436 | -0.2 (0.67) | -0.3 (0.65)
  Week 4, n=216, 427 | -0.3 (0.72) | -0.4 (0.84)
  Week 6, n=196, 418 | -0.4 (0.78) | -0.4 (0.80)
  Week 8, n=189, 413 | -0.4 (0.89) | -0.6 (0.92)
  Week 12, n=164, 401 | -0.5 (1.11) | -0.8 (1.09)
  Week 16, n=138, 375 | -0.7 (1.10) | -1.0 (1.14)
  Week 20, n=134, 362 | -0.7 (1.24) | -1.2 (1.27)
  Week 24, n=87, 248 | -0.6 (1.19) | -1.5 (1.42)
  Week 28, n=73, 201 | -0.9 (1.63) | -1.6 (1.42)
  Week 32, n=68, 183 | -0.7 (1.25) | -1.5 (1.46)
  Week 36, n=67, 174 | -0.7 (1.30) | -1.6 (1.51)
  Week 40, n=63, 169 | -0.7 (1.42) | -1.6 (1.59)
  Week 44, n=64, 166 | -0.8 (1.53) | -1.7 (1.61)
  End of Treatment, n=212, 416 | -0.7 (1.33) | -1.5 (1.66)
  4-week FU, n=202, 402 | -0.7 (1.37) | -1.3 (1.66)
  12-week FU, n=196, 398 | -0.5 (1.54) | -1.0 (1.79)
  24-week FU, n=195, 390 | -0.3 (1.81) | -0.6 (1.78)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported for the Double-blind (DB) on-treatment + 30 days period (up to Study Week 72).
Description: In the study, AEs were collected during the Open-Label (OL) Pre-Antiviral Treatment Phase and the Double-Blind (DB) Phase, which included antiviral therapy and a 6-month post-therapy follow-up. Data for SAEs and AEs are presented for the Safety Population, comprised of all randomized participants who received the study drug.
Arm/Group | Eltrombopag: OL Phase | Placebo+Antiviral Therapy: DB Phase | Eltrombopag+Antiviral Therapy: DB Phase
Serious Adverse Events (participants affected / at risk) | 8/715 | 35/232 | 89/449
Other Adverse Events (participants affected / at risk) | 49/715 | 219/232 | 424/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag: OL Phase (N=715) | Placebo+Antiviral Therapy: DB Phase (N=232) | Eltrombopag+Antiviral Therapy: DB Phase (N=449)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 1
Oesophageal Varices Hemorrhage (Gastrointestinal disorders) | 1 | 2 | 7
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 6
Pyrexia (General disorders) | 1 | 0 | 3
Pneumonia (Infections and infestations) | 1 | 2 | 4
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 3 | 4
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 4
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Gastric Varices Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 4
Peritonitis Bacterial (Infections and infestations) | 0 | 2 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3
Abscess Limb (Infections and infestations) | 0 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 2
Septic Shock (Infections and infestations) | 0 | 0 | 2
Bacteremia (Infections and infestations) | 0 | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Diarrhea Infectious (Infections and infestations) | 0 | 0 | 1
Disseminated Tuberculosis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Meningitis Cryptococcal (Infections and infestations) | 0 | 0 | 1
Prostatic Abscess (Infections and infestations) | 0 | 0 | 1
Renal Abscess (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Acinetobacter Bacteremia (Infections and infestations) | 0 | 1 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Hemolytic Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1 | 7
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis Alcoholic (Hepatobiliary disorders) | 0 | 0 | 1
Hepatorenal Syndrome (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 1
Edema Peripheral (General disorders) | 0 | 0 | 1
Multi-organ Failure (General disorders) | 0 | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 4
Encephalopathy (Nervous system disorders) | 0 | 0 | 2
Brain Edema (Nervous system disorders) | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Vocal Cord Paralysis (Nervous system disorders) | 0 | 0 | 1
Ruptured Cerebral Aneurysm (Nervous system disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 2 | 2
Cataract Nuclear (Eye disorders) | 0 | 0 | 1
Eye Disorder (Eye disorders) | 0 | 0 | 1
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 2
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 2
Cystitis Ulcerative (Renal and urinary disorders) | 0 | 0 | 1
Urethral Polyp (Renal and urinary disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea Exertional (Reproductive system and breast disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Pleuropericarditis (Cardiac disorders) | 0 | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Retinal Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bleeding Varicose Vein (Vascular disorders) | 0 | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 1
Varicose Vein (Vascular disorders) | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1
Transaminases Increased (Investigations) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Juvenile Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 2
Epidermolysis Bullosa (Congenital, familial and genetic disorders) | 0 | 1 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Alcohol Use (Social circumstances) | 0 | 0 | 1
Portal Shunt (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag: OL Phase (N=715) | Placebo+Antiviral Therapy: DB Phase (N=232) | Eltrombopag+Antiviral Therapy: DB Phase (N=449)
Headache (Nervous system disorders) | 49 | 47 | 107
Neutropenia (Blood and lymphatic system disorders) | 0 | 95 | 170
Anemia (Blood and lymphatic system disorders) | 0 | 78 | 183
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 85 | 69
Leukopenia (Blood and lymphatic system disorders) | 0 | 39 | 70
Fatigue (General disorders) | 0 | 60 | 139
Pyrexia (General disorders) | 0 | 53 | 139
Influenza Like Illness (General disorders) | 0 | 40 | 70
Asthenia (General disorders) | 0 | 34 | 66
Edema Peripheral (General disorders) | 0 | 20 | 56
Chills (General disorders) | 0 | 12 | 58
Irritability (General disorders) | 0 | 17 | 46
Nausea (Gastrointestinal disorders) | 0 | 30 | 86
Diarrhea (Gastrointestinal disorders) | 0 | 27 | 82
Vomiting (Gastrointestinal disorders) | 0 | 17 | 31
Abdominal Pain (Gastrointestinal disorders) | 0 | 12 | 33
Dyspepsia (Gastrointestinal disorders) | 0 | 16 | 27
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 11 | 29
Ascites (Gastrointestinal disorders) | 0 | 7 | 32
Constipation (Gastrointestinal disorders) | 0 | 11 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 34 | 77
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 33 | 30
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 15 | 38
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 28
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 30
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 27 | 68
Rash (Skin and subcutaneous tissue disorders) | 0 | 24 | 49
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 15 | 50
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 14 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 26 | 65
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 17 | 55
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 15 | 46
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 10 | 26
Dizziness (Nervous system disorders) | 0 | 24 | 26
Insomnia (Psychiatric disorders) | 0 | 44 | 79
Depression (Psychiatric disorders) | 0 | 11 | 38
Anxiety (Psychiatric disorders) | 0 | 13 | 18
Blood Bilirubin Increased (Investigations) | 0 | 8 | 44
White Blood Cell Count Decreased (Investigations) | 0 | 9 | 32
Hemoglobin Decreased (Investigations) | 0 | 9 | 31
Weight Decreased (Investigations) | 0 | 9 | 25
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 30 | 78
Urinary Tract Infection (Infections and infestations) | 0 | 8 | 39
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 12 | 24
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 5 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.